CLINICAL TRIAL: NCT03979820
Title: A Phase I Parallel Group Study in Healthy Subjects to Evaluate the Effect of Multiple Oral Doses of BI 1467335 and Phenelzine as Positive Control on Blood Pressure Response to Oral Tyramine (Double-blind, Randomised, Placebo-controlled Design for BI 1467335 Treatment Groups, Open Label for Phenelzine)
Brief Title: A Study in Healthy People to Test How Combining BI 1467335 and Tyramine Affects Blood Pressure
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study discontinued - testing of highest dose obsolete
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1386.16; 2018-003965-32 (EudraCT Number)
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Phenelzine; Tyramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 10 mg BI 1467335/10 mg BI 1467335 + Tyramine (Experimental)
  Interventions: Drug: BI 1467335; Drug: Tyramine
- 15 mg BI 1467335/15 mg BI 1467335 + Tyramine (Experimental)
  Interventions: Drug: BI 1467335; Drug: Tyramine
- Phenelzine/Phenelzine + Tyramine (Active Comparator)
  Interventions: Drug: Phenelzine sulfate; Drug: Tyramine
- Placebo/Placebo + Tyramine (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Tyramine

INTERVENTIONS:
Drug: BI 1467335 — Film-coated tablet
  Arms: 10 mg BI 1467335/10 mg BI 1467335 + Tyramine; 15 mg BI 1467335/15 mg BI 1467335 + Tyramine
Drug: Placebo — Film-coated tablet
  Arms: Placebo/Placebo + Tyramine
Drug: Phenelzine sulfate — Film-coated tablet
  Arms: Phenelzine/Phenelzine + Tyramine
Drug: Tyramine — Capsules

SUMMARY:
The main objective of the study is investigate the effect of escalating doses of oral tyramine on systolic blood pressure (SBP) at baseline and following an oral treatment with BI 1467335 up to 39 days at a low or high dose once daily compared to placebo and phenelzine (Nardil®) as positive control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device (in case of oral contraceptives start of contraception at least 30 days before administration of trial medication)
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
* Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of FSH above 33,4 U/L and estradiol below 71,6 pmol/L is confirmatory) Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Use of monoamine oxidase (MAO) inhibitors within 90 days before tyramine dosing
* Use of fluoxetine within 5 weeks before tyramine dosing
* Use of over-the-counter sympathomimetic or grapefruit products within 7 days before tyramine dosing
* Subject has a known intolerability to tyramine-containing foods
* At screening, no increase of systolic blood pressure > 30 mmHg during tyramine challenge at the highest tested dose of 700 mg tyramine

Female subjects will not be allowed to participate, if any of the following apply:

* Positive pregnancy test, pregnancy, or plans to become pregnant within 30 days after study completion
* Lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a a randomised, double-blind, placebo controlled clinical trial in healthy subjects to evaluate the effects of multiple oral doses of BI 1467335 and phenelzine as positive control on blood pressure response to oral tyramine.
  Trial was ended prematurely due to lockdown of the trial site by the Covid-19 pandemic.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct.
Groups:
- Placebo/Placebo + Tyramine: Tyramine was administered during the screening process (tyramine screening/baseline challenge, Day -11 to Day -2) and at steady state (tyramine steady state challenge, Day 29 up to Day 39) following multiple doses of placebo matching BI 1467335. During tyramine baseline challenge and tyramine steady state challenge participants received escalating tyramine doses until tyramine dose caused an increase of systolic blood pressure (SBP) ≥ 30 millimetre of mercury (mmHg) for at least 3 consecutive measurements (TYR30). During the tyramine baseline challenge the planned tyramine doses were 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 milligram (mg) once daily orally with 240 milliliter (ml) of water. During the tyramine steady state challenge the planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg once daily orally with 240 ml of water. 2 or 3 film-coated tablets of 5 mg of placebo matching BI 1467335 were administered once daily (daily dosage: 10 or 15 mg) orally with 240 ml of water from Day 1 up to Day 39. Treatment with placebo matching BI 1467335 was to be stopped as soon as the individual participant had attained TYR30 on treatment.
- Phenelzine/Phenelzine + Tyramine: Tyramine was administered during the screening process (tyramine screening/baseline challenge, Day -11 to Day -2) and at steady state (tyramine steady state challenge, Day 8 to Day 19) following multiple doses of phenelzine sulfate (Nardil®). During tyramine baseline challenge and tyramine steady state challenge participants received escalating tyramine doses until tyramine dose caused an increase of systolic blood pressure (SBP) ≥ 30 millimetre of mercury (mmHg) for at least 3 consecutive measurements (TYR30). During the tyramine baseline challenge the planned tyramine doses were 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 milligram (mg) once daily orally with 240 milliliter (ml) of water. During the tyramine steady state challenge the planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg once daily orally with 240 ml of water. Additionally an intermediate tyramine dose of 150 mg once daily was administered. 1 film-coated tablet of 15 mg of phenelzine sulfate was administered twice daily (daily dosage: 30 mg) from Day 1 to Day 18 and once daily (daily dosage: 15 mg) on Day 19 orally with 240 ml of water. Treatment with phenelzine sulfate was stopped as soon as the individual participant attained TYR30 on treatment.
- 10 mg BI 1467335/10 mg BI 1467335 + Tyramine: Tyramine was administered during the screening process (tyramine screening/baseline challenge, Day -11 to Day -2) and at steady state (tyramine steady state challenge, Day 29 up to Day 39) following multiple doses of BI 1467335. During tyramine baseline challenge and tyramine steady state challenge participants received escalating tyramine doses until tyramine dose caused an increase of systolic blood pressure (SBP) ≥ 30 millimetre of mercury (mmHg) for at least 3 consecutive measurements (TYR30). During the tyramine baseline challenge the planned tyramine doses were 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 milligram (mg) once daily orally with 240 milliliter (ml) of water. During the tyramine steady state challenge the planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg once daily orally with 240 ml of water. 2 film-coated tablets of 5 mg of BI 1467335 were administered once daily (daily dosage: 10 mg) orally with 240 ml of water from Day 1 up to Day 39. Treatment with BI 1467335 was stopped as soon as the individual participant attained TYR30 on treatment.
- 15 mg BI 1467335/15 mg BI 1467335 + Tyramine: Tyramine was administered during the screening process (tyramine screening/baseline challenge, Day -11 to Day -2) and at steady state (tyramine steady state challenge, Day 29 up to Day 39) following multiple doses of BI 1467335. Participants received escalating tyramine doses until tyramine dose caused an increase of systolic blood pressure (SBP) ≥ 30 millimetre of mercury (mmHg) for at least 3 consecutive measurements (TYR30). During the tyramine baseline challenge the planned tyramine doses were 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 milligram (mg) once daily orally with 240 milliliter (ml) of water. During the tyramine steady state challenge the planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg once daily orally with 240 ml of water. 3 film-coated tablets of 5 mg of BI 1467335 were administered once daily (daily dosage: 15 mg) orally with 240 ml of water from Day 1 up to Day 39. Treatment with BI 1467335 was to be stopped as soon as the individual participant attained TYR30 on treatment.
Period: Overall Study
Arm/Group | Placebo/Placebo + Tyramine | Phenelzine/Phenelzine + Tyramine | 10 mg BI 1467335/10 mg BI 1467335 + Tyramine | 15 mg BI 1467335/15 mg BI 1467335 + Tyramine
Started | 13 | 14 | 16 | 10
Completed | 7 | 14 | 15 | 0
Not Completed | 6 | 0 | 1 | 10
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Permanent discontinuation of the trial due to Covid-19 pandemic | 5 | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This analysis set included all subjects who were randomised and received at least one dose of trial medication. The TS was used for the analysis of safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Placebo + Tyramine | Phenelzine/Phenelzine + Tyramine | 10 mg BI 1467335/10 mg BI 1467335 + Tyramine | 15 mg BI 1467335/15 mg BI 1467335 + Tyramine | Total
Number analyzed (Participants) | 13 | 14 | 16 | 10 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (8.1) | 31.4 (8.6) | 30.9 (6.8) | 30.4 (8.6) | 31.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 7 | 3 | 21
  Male | 8 | 8 | 9 | 7 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 12 | 14 | 15 | 9 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 1 | 3
  Asian | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 12 | 11 | 12 | 7 | 42
  More than one race | 0 | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Tyramine dose at baseline to reach TYR30 [Mean (Standard Deviation); unit: Milligramm (mg)] — Tyramine dose at baseline to reach TYR30 is the dose of tyramine during the baseline tyramine challenge (from Day -11 up to Day-2) causing an increase of systolic blood pressure (SBP)≥30 millimetre of mercury (mmHg) in at least 3 consecutive measurements (TYR30).
  Milligramm (mg) | 453.846 (133.012) | 464.286 (121.574) | 456.250 (126.326) | 390.000 (159.513) | 445.283 (132.384)

OUTCOME MEASURES:

1. Primary Outcome: Tyramine Sensitivity Factor (TSF)
Description: TSF was defined as ratio of the tyramine dose causing an increase of systolic blood pressure (SBP) ≥ 30 millimetre of mercury (mmHg) for at least 3 consecutive measurements (TYR30) at baseline and at steady state of BI 1467335, placebo or phenelzine. Geometric Mean is the Geometric Least Squares Mean and is extracted from the ANOVA model that includes all treatments. Standard error is the geometric standard error of the mean (gSE) and is extracted from the ANOVA model that includes all treatments.
Time Frame: At baseline (Day -11 up to Day-2) and at steady state (Day 29 up to Day 39 for the "Placebo/Placebo + Tyramine" and "10 mg BI 1467335/10 mg BI 1467335 + Tyramine" arms, Day 8 up to Day 19 for the "Phenelzine/ Phenelzine + Tyramine" arm).
Population: Per protocol analysis set (PPS): This analysis set included all participants in the TS who provided at least one endpoint that was defined as primary and was not excluded due to a protocol violation relevant. Descriptive and model-based analyses of the primary endpoint were based on the PPS. Participants of the arms "15 mg BI 1467335/15 mg BI 1467335 + Tyramine" and "Placebo/Placebo + Tyramine" who could not complete the tyramine steady state challenge were excluded from the analysis.
Measure: Geometric Least Squares Mean (Standard Error); unit: Ratio of tyramine dose
Arm/Group | Placebo/Placebo + Tyramine | Phenelzine/Phenelzine + Tyramine | 10 mg BI 1467335/10 mg BI 1467335 + Tyramine
Number analyzed (Participants) | 7 | 14 | 14
Ratio of tyramine dose | 0.98 (1.25) | 5.31 (1.17) | 1.20 (1.17)
Statistical Analysis 1: Comparison: Placebo/Placebo + Tyramine vs Phenelzine/Phenelzine + Tyramine; The statistical model used for the analysis of the primary endpoint was an analysis of variance (ANOVA) model on the logarithmic scale for each treatment relative to placebo. TSF was log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the fixed effects 'treatment'; Test type: Other; ANOVA; Ratio of geometric mean TSFs = 544.36, 90% CI 2-sided [340.57 to 870.09], Standard Error of Mean 1.32 — The arm "Phenelzine/Phenelzine + Tyramine" represented the numerator. The arm "Placebo/Placebo + Tyramine" represented the denominator
Statistical Analysis 2: Comparison: Placebo/Placebo + Tyramine vs 10 mg BI 1467335/10 mg BI 1467335 + Tyramine; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of geometric mean TSFs = 123.22, 90% CI 2-sided [77.09 to 196.95], Standard Error of Mean 1.32 — The arm "10 mg BI 1467335/10 mg BI 1467335 + Tyramine" represented the numerator. The arm "Placebo/Placebo + Tyramine" represented the denominator

ADVERSE EVENTS:
Time Frame: Tyramine screening: From Day -11 to time of first administration of BI 1467335, placebo or phenelzine Day 1, up to 11 days. Placebo, 10 mg BI 1467335, 15 mg BI 1467335: From Day 1 to Day 29, up to 28 days. Phenelzine: From Day 1 to Day 8, up to 7 days. Placebo + Tyramine, 10 mg BI 1467335 + Tyramine, 15 mg BI 1467335 + Tyramine: From Day 29 up to End of trial (EoT), up to 23 days. Phenelzine +Tyramine: From Day 8 until EoT, up to 24 days.
Description: Treated set (TS): This analysis set included all subjects who were randomised and received at least one dose of trial medication.
Groups:
- Tyramine Screening: As part of the screening procedure, participants were challenged (tyramine screening/baseline challenge) from Day -11 up to Day -2 with escalating oral doses of tyramine. Planned tyramine doses were 10, 25, 50, 100, 200, 300, 400, 500, 600, 700 mg given once daily orally with 240 ml of water. In each individual participant, the tyramine dose escalation was stopped when SBP increased ≥30 mmHg in at least 3 consecutive measurements (TYR30). Participants who did not attain the predefined systolic BP target elevation within 4 h after 700 mg tyramine were not to be included in the trial.
- Placebo: From Day 1 to Day 28 participants received once daily 2 or 3 film-coated tablets of 5 mg of placebo matching BI 1467335 administered once daily (daily dosage: 10 or 15 mg) orally with 240 ml of water.
- Phenelzine: From Day 1 to Day 7 participants received 1 film-coated tablet of 15 mg of phenelzine sulfate administered twice daily (daily dosage: 30 mg) orally with 240 ml of water.
- 10 mg BI 1467335: From Day 1 to Day 28 participants received 2 film-coated tablets of 5 mg of BI 1467335 administered once daily (daily dosage:10 mg) orally with 240 ml of water.
- 15 mg BI 1467335: From Day 1 to Day 28 participants received 3 film-coated tablets of 5mg of BI 1467335 administered once daily (daily dosage: 15 mg) orally with 240 ml of water.
- Placebo + Tyramine: Participants received from Day 29 up to Day 39 concomitant medication of 2 0r 3 film-coated tablets of 5 mg of placebo matching BI 1467335 administered once daily (daily dosage:10 or 15mg) orally with 240 ml of water and escalating doses of tyramine (tyramine steady state challenge) until TYR30 was reached. The planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg given once daily orally with 240 ml of water. Treatment with placebo matching BI 1467335 was to be stopped as soon as the individual subject had attained TYR30 on treatment.
- Phenelzine + Tyramine: Participants received from Day 8 up to Day 19 concomitant medication of 1 film-coated tablets of 15 mg of phenelzine sulfate (Nardil®) administered twice daily from Day 8 up to Day 18 (daily dosage: 30 mg) and once daily on Day 19 (daily dosage: 15 mg) orally with 240 ml of water and escalating doses of tyramine (tyramine steady state challenge) until TYR30 was reached. The planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg given once daily orally with 240 ml of water. Additionally an intermediate tyramine dose of 150 mg once daily was administered. Treatment with phenelzine sulfate was stopped as soon as the individual subject attained TYR30 on treatment.
- 10 mg BI 1467335 + Tyramine: Participants received from Day 29 up to Day 39 concomitant medication of 2 film-coated tablets of 5mg of BI 1467335 administered once daily (total dosage: 10 mg) orally with 240 ml of water and escalating doses of tyramine (tyramine steady state challenge) until TYR30 was reached. The planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg given once daily orally with 240 ml of water. Treatment with BI 1467335 was stopped as soon as the individual subject attained TYR30 on treatment.
- 15 mg BI 1467335 + Tyramine: Participants received from Day 29 up to Day 39 concomitant medication of 3 film-coated tablets of 5 mg of BI 1467335 administered once daily (daily dosage 15mg) orally with 240 ml of water and escalating doses of tyramine (tyramine steady state challenge) until TYR30 was reached. The planned tyramine doses were 5, 10, 25, 50, 100, 200, 300, 400, 500, 600, and 700 mg given once daily orally with 240 ml of water. Treatment with BI 1467335 was to be stopped as soon as the individual subject had attained TYR30 on treatment.
Arm/Group | Tyramine Screening | Placebo | Phenelzine | 10 mg BI 1467335 | 15 mg BI 1467335 | Placebo + Tyramine | Phenelzine + Tyramine | 10 mg BI 1467335 + Tyramine | 15 mg BI 1467335 + Tyramine
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/13 | 0/14 | 0/16 | 0/10 | 0/9 | 0/14 | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/13 | 0/14 | 0/16 | 0/10 | 0/9 | 0/14 | 1/15 | 0/6
Other Adverse Events (participants affected / at risk) | 39/53 | 9/13 | 11/14 | 8/16 | 7/10 | 8/9 | 14/14 | 10/15 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tyramine Screening (N=53) | Placebo (N=13) | Phenelzine (N=14) | 10 mg BI 1467335 (N=16) | 15 mg BI 1467335 (N=10) | Placebo + Tyramine (N=9) | Phenelzine + Tyramine (N=14) | 10 mg BI 1467335 + Tyramine (N=15) | 15 mg BI 1467335 + Tyramine (N=6)
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tyramine Screening (N=53) | Placebo (N=13) | Phenelzine (N=14) | 10 mg BI 1467335 (N=16) | 15 mg BI 1467335 (N=10) | Placebo + Tyramine (N=9) | Phenelzine + Tyramine (N=14) | 10 mg BI 1467335 + Tyramine (N=15) | 15 mg BI 1467335 + Tyramine (N=6)
Nausea (Gastrointestinal disorders) | 13 | 2 | 0 | 1 | 0 | 2 | 9 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 0 | 2 | 0 | 0 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 1 | 5 | 2 | 1 | 0 | 4 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 2
Catheter site related reaction (General disorders) | 0 | 2 | 2 | 1 | 0 | 2 | 1 | 2 | 0
Chest discomfort (General disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Medical device site irritation (General disorders) | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Medical device site dermatitis (General disorders) | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Medical device site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 20 | 3 | 1 | 4 | 4 | 2 | 6 | 4 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 18 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Fear (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laziness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The sponsor decided to permanently discontinue the trial on 14 April 2020 due to lock down of the trial site enforced by the Covid-19 pandemic. Therefore some of the planned analysis were not performed due to lack of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT03979820/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03979820/SAP_001.pdf